CLINICAL TRIAL: NCT04921033
Title: Exclusive Enteral Nutrition in Patients With Ileocaecal Crohn's Disease (XENIC): an Open-label, Multicenter, Prospective, Randomized Clinical Trial
Brief Title: Exclusive Enteral Nutrition in Patients With Ileocaecal Crohn's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Salih Tokmak, Asistant Professor, Duzce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EEN in ileocaecal Crohn's
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease; Nutrient; Excess; Remission/Regression
Keywords: enteral nutrition; induction of remission; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide; Prednisolone; Methylprednisolone; Azathioprine

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, multicenter, interventional, parallel-group study, designed to evaluate the efficacy and tolerability of EEN in inducing clinical remission at 12 weeks in subjects with ileocaecal CD.
  Patients will receive EEN for 8 weeks, initially building up to the full required volume of formula over the first 3 to 4 days, depending on tolerance and side effects After the completion of the period of EEN, foods will be reintroduced slowly and supplementary enteral nutrition will be continued for another 4 weeks.
  A total of 256 patients with ileocaecal CD will be randomized in a 1:1 ratio to receive steroids and EEN. Each of the treatment arms will comprise 128 subjects. In order to make the groups comparable, randomization will be stratified according to the severity of the disease according to Crohn's Disease Activity Index (CDAI):
  1. CDAI between 150-220 --> Mild
  2. CDAI between 220-450 --> Moderate
  3. CDAI>450 --> Severe
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exclusive Enteral Nutrition (Experimental): 35kcal/kg/day EEN (Nestle Modulen®) - Subjects will take medicine and EEN solution orally themselves.
  Interventions: Dietary Supplement: EEN (Nestle Modulen®)
- Standard of care (Active Comparator): * Budesonide 9mg/day for mild disease
  * Prednisolone 1mg/kg, maximum 40mg/day in decreasing doses (40mg for 4 weeks followed by a fixed taper for 6 weeks) for moderate-to-severe disease for 12 weeks.
  * Patients with moderate-to-severe disease in the steroid group will also receive 2mg/kg azathioprine. The dose of azathioprine will be adjusted according to abnormalities of white blood cell (WBC) count, platelet count, liver function tests (LFTs; i.e. alanine transaminase [ALT], aspartate transaminase [AST], alkaline phosphatase), lipase, blood urea nitrogen (BUN), and serum creatinine.
  Interventions: Drug: Standart of care

INTERVENTIONS:
Dietary Supplement: EEN (Nestle Modulen®) — 35kcal/kg/day for every patient
  Arms: Exclusive Enteral Nutrition
Drug: Standart of care — * Budesonide 9mg/day for mild disease
  * Prednisolone 1mg/kg, maximum 40mg/day in decreasing doses (40mg for 4 weeks followed by a fixed taper for 6 weeks) for moderate-to-severe disease for 12 weeks.
  * Patients with moderate to severe disease in the steroid group will also receive 2mg/kg azathioprine. The dose of azathioprine will be adjusted according to abnormalities of white blood cell (WBC) count, platelet count, liver function tests (LFTs; i.e. alanine transaminase [ALT], aspartate transaminase [AST], alkaline phosphatase), lipase, blood urea nitrogen (BUN), and serum creatinine.
  Other Names: Budesonide (Budenofalk®), Prednisolone (Deltacortril®), Azathioprine (Imuran®)
  Arms: Standard of care

SUMMARY:
Inflammatory bowel diseases are chronic and progressive entities, triggered by exposure to environmental factors in individuals with a genetic background.

One of the most common environmental factors is the type of diet which is a key influencer on pathogenesis. Nutrients alter the intestinal microbiota, thus changing the intestinal permeability. The Western-type diet encompasses sugar, fat, and protein-rich products that have some deleterious effects on the intestinal microbiome compared to the plant-based Mediterranean-type diet.

Based on this fact, diet-based therapeutic efforts have been used extensively in pediatric Crohn's disease patients and there is strong evidence that exclusive enteral nutrition (EEN) is as effective as corticosteroids to induce both clinical and endoscopic remission but this treatment strategy is underutilized in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged between 18-75 years with a diagnosis of ileocolonic Crohn's disease (CD) confirmed using endoscopy and/or imaging technology at most 3 months prior.
* Participant or his/her legal representative have voluntarily signed and dated an informed consent approved by and compliant with the requirements of this study protocol which has been approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) Adequate cardiac, renal, and hepatic function as determined by the Principal Investigator and demonstrated by Screening laboratory evaluations, questionnaires, and physical examination results that do not indicate an abnormal clinical condition that would place the participant at undue risk preclude participation in the study.
* Participant must be able to orally administer study medication/nutrient or have a designee or Healthcare Professional who can assist

Exclusion Criteria:

* Previous or current use of any medication for Crohn's disease such as biologics, immunomodulators (e.g., methotrexate, azathioprine, 6-mercaptopurine, JAK inhibitor, alpha-integrin), and corticosteroids
* Presence of complications (Fistula, abscess, fibrotic disease, imminent risk of surgery)
* Participants with a poorly controlled medical condition such as uncontrolled diabetes with a documented history of recurrent infections, unstable ischemic heart disease, moderate to severe congestive heart failure (New York Heart Association [NYHA] class III or IV), recent cerebrovascular accident, and any other condition which, in the opinion of the Investigator or the sponsor, would put the participant at risk by participation in the protocol
* Participants with positive C. difficile stool assay at screening.
* Rescue therapy with steroids, depending on the severity of the disease will be initiated for patients in the EEN group who do not respond clinically and will be excluded from the study. If the number of clinically unresponsive patients was greater than 25% of the total EEN population, the study will be stopped. Criteria for clinical response are described in the "Outcome Measures" section.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with mucosal healing | 12 weeks
  Defined as Simple Endoscopic Score for Crohn's Disease (SES-CD) ≤2, at 12 weeks after randomization. The ileocolonoscopies will be evaluated by the site.
  SES-CD is an index for determining the severity of Crohn's disease. The SES-CD considers size of ulcerations, ulcerated surface, effected surface and the presence of narrowings, evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). The score ranges from 0 to 60 where higher scores indicate more severe endoscopic activity.
Percentage of patients that tolerate the EEN by week 12 | 12 weeks
  Defined as withdrawal from the study from randomization through 12 weeks after randomization

SECONDARY OUTCOMES:
Endoscopic response | 12 weeks
  Defined as decrease in SES-CD > 50% from baseline at 12 weeks after randomization
Mean change from baseline in SES-CD at 12 weeks after randomization | 12 weeks
  Mean change from baseline in SES-CD
Mean change from baseline in CDAI over time (Time Frame: Baseline, 4, 8 and 12 weeks after randomization) | 12 weeks
  The Crohn's Disease Activity Index (CDAI) is a research tool used to quantify the symptoms of patients with Crohn's disease. Participants were asked to record the frequency of stools, abdominal pain and general well-being on a daily basis. In addition to the diary data, the investigator assessed the following for the calculation of CDAI: presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. The CDAI is the sum of the products of each item multiplied by a weighting factor and generally ranges from 0 up to 600, where remission of Crohn's disease is defined as CDAI < 150, and severe disease is defined as CDAI > 450. A negative change from baseline indicates improvement.
Time to clinical remission (Time frame: from randomization through 12 weeks after randomization) | 12 weeks
  Clinical remission was defined as:
  * CDAI < 150
  * PRO-2 abdominal pain (AP) score≤1 (7 day average) and liquid/very soft stool frequency (SF) score≤3 (7 day average)
  Two-item Patient Reported Outcome (PRO-2) is a health outcome directly reported by the patient to quantify a treatment's efficacy that is derived from CDAI diary card. Participants were asked to record daily number of liquid or very soft stools and the severity of abdominal pain (defined as; 0=none, 1=mild, 2=moderate 3=severe). PRO-2 is the sum of the products of each item multiplied by a weighing factor. PRO-2 scores that correspond to CDAI thresholds are:
  Mild Moderate Severe CDAI 150 220 450 PRO-2 8 14 34
Time to clinical response (Time frame: from randomization through 12 weeks after randomization) | 12 weeks
  Clinical response was defined as:
  * CDAI reduction ≥100 from baseline
  * PRO-2 reduction ≥8 from baseline
Mean change from baseline in C-reactive protein (CRP) over time (Time Frame: 4, 8 and 12 weeks after randomization) | 12 weeks
  Changes in CRP levels
Mean change from baseline in fecal calprotectin (FC) over time (Time Frame: 4, 8 and 12 weeks after randomization) | 12 weeks
  Changes in fecal calprotectin levels
Mean change from baseline in PRO-2 (Time Frame: Baseline and 12 weeks after randomization) | 12 weeks
  Two-item Patient Reported Outcome (PRO-2) is a health outcome directly reported by the patient to quantify a treatment's efficacy that is derived from CDAI diary card. Participants were asked to record daily number of liquid or very soft stools and the severtiy of abdominal pain (defined as; 0=none, 1=mild, 2=moderate 3=severe). PRO-2 is the sum of the products of each item multiplied by a weighing factor. PRO-2 scores that correspond to CDAI thresholds are:
  Mild Moderate Severe CDAI 150 220 450 PRO-2 8 14 34
Change from baseline in SIBDQ total score (Time Frame: Baseline and 12 weeks after randomization) | 12 weeks
  Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a 10-item HrQOL questionnaire designed to quantify the changes in patients' daily activity, related to Crohn's disease symptoms. Participants were asked questions about physical, social, emotional, and systemic aspects and scored on a 7-point scale from 1 (severe problem) to 7 (no problems at all). The score ranges from 1 to 70 where higher scores indicate better HrQOL.
Change in Robarts Histopathology Index (RHI) (Time Frame: Baseline and 12 weeks after randomization) | 12 weeks
  RHI is a research tool used to quantify the histologic changes and to assess the degree of inflammation in the mucosa.
  RHI= 1xchronic inflammatory infiltrate level (4 levels)
  * 2 x lamina propria neutrophils (4 levels)
  * 3 x neutrophils in epithelium (4 levels)
  * 5 x erosion or ulceration (4 levels)
  The total score ranges from 0 (no disease activity) to 33 (severe disease activity). RHI≤3 corresponds to histologic remission.
Number of Crohn's disease-related hospitalizations after randomization (Time Frame: From randomization through 12 weeks after randomization) | 12 weeks
  Hospitalization was defined as a visit to hospital/clinic resulting in admission and overnight stay in hospital/clinic. Hospitalization due to emergency was defined as a hospitalization admitted through the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Salih Tokmak, Principal Investigator — Duzce University
Locations (1):
- Duzce University School of Medicine, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR) will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication, for a year